CLINICAL TRIAL: NCT05685836
Title: 89Zr-Bevacizumab PET/CT Imaging of Vestibular Schwannomas for the Prediction of Bevacizumab Treatment Effect in Patients With Symptomatic Neurofibromatosis Type 2
Brief Title: 89Zr-Bevacizumab PET/CT Imaging in NF2 Patients
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Hans Gelderblom, Prof. A.J. Gelderblom, MD, PhD, Head of Medical Oncology, Principal Investigator, Leiden University Medical Center
Other Study IDs: NF2PET; 2020-000156-35 (EudraCT Number)
Record Dates: First submitted 2022-12-05; First posted 2023-01-17 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Neurofibromatosis 2
Keywords: neurofibromatosis 2; NF2-related schwannomatosis; vestibular schwannoma; bevacizumab; 89Zr-Bevacizumab; PET/CT imaging; hearing
MeSH Terms: conditions — Neurofibromatosis 2; Neuroma, Acoustic | interventions — 89Zr-bevacizumab; Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Bevacizumab: After determining eligibility, all patients will undergo standard-of-care treatment with the sole addition of a pre-treatment 89Zr-Bevacizumab PET/CT-scan. Patients will first receive 5 mg 89Zr-Bevacizumab 4 days before PET/CT scan. This is followed by standard-of-care intravenous 7.5mg/kg bevacizumab (Avastin) therapy, administered every three weeks for six months
  Interventions: Drug: Bevacizumab Zirconium Zr-89

INTERVENTIONS:
Drug: Bevacizumab Zirconium Zr-89 — See Arm description.
  Other Names: Avastin; 89Zr-Bevacizumab; Bevacizumab

SUMMARY:
Bevacizumab can be an effective treatment for individuals with NF2 and improve different nerve functions (like hearing, tinnitus or balance problems) and the quality of life of NF2 patients. However, bevacizumab is not effective in all patients or all tumors, at the cost of moderate toxicity and considerable financial burden.

Therefore, this observational study will validate an imaging biomarker method to predict bevacizumab efficacy in order to avoid adverse effects and high costs in non-responders to bevacizumab treatment. Patients will undergo standard-of-care treatment with the sole addition of a pre-treatment 89Zr-Bevacizumab PET/CT-scan. Per standard-of-care bevacizumab therapy is administered every three weeks for six months. To monitor treatment effect, follow-up is performed at 3-month intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Confirmed diagnosis of NF2 by revised Manchester criteria
* Provided written informed consent
* Patients must have measurable disease, defined as at least one VS > 0.4 ml (on volumetric analysis) that can be accurately measured by contrast-enhanced T1-weighted cranial MRI scan.
* Eligible and planned for bevacizumab treatment

Exclusion Criteria:

* Patients with a contra-indication for PET and MRI, such as pregnancy and metal elements.
* Patients with a known allergy to substances used in this study
* Concurrent treatment with Everolimus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a confirmed diagnosis of NF2 and candidate for bevacizumab therapy.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Hearing response (HR) - WRS | Baseline
  Word Recognition Score (WRS), % at x dB
Hearing response (HR) - WRS | 3 months
  Word Recognition Score (WRS), % at x dB
Hearing response (HR) - WRS | 6 months
  Word Recognition Score (WRS), % at x dB
Hearing response (HR) - PTA | Baseline
  Pure Tone Average (PTA), in dB
Hearing response (HR) - PTA | 3 months
  Pure Tone Average (PTA), in dB
Hearing response (HR) - PTA | 6 months
  Pure Tone Average (PTA), in dB
Radiographic response (RR) - tumor volumetry on MRI | Baseline
  Size change in volumetric MRI (REiNS criteria); volumetry in mL or mm
Radiographic response (RR) - tumor volumetry on MRI | 3 months
  Size change in volumetric MRI (REiNS criteria); volumetry in mL or mm
Radiographic response (RR) - tumor volumetry on MRI | 6 months
  Size change in volumetric MRI (REiNS criteria); volumetry in mL or mm
Radiographic response (RR) - ADC | Baseline
  Apparent diffusion coefficient (ADC) of tumor of interest, in mm2/s, on greatest diameter
Radiographic response (RR) - ADC | 3 months
  Apparent diffusion coefficient (ADC) of tumor of interest, in mm2/s, on greatest diameter
Radiographic response (RR) - ADC | 6 months
  Apparent diffusion coefficient (ADC) of tumor of interest, in mm2/s, on greatest diameter
Radiographic response (RR) - Microbleeds | Baseline
  Location and number of microbleeds
Radiographic response (RR) - Microbleeds | 3 months
  Location and number of microbleeds
Radiographic response (RR) - Microbleeds | 6 months
  Location and number of microbleeds
Radiographic response (RR) - Diffusion restriction | Baseline
  Diffusion restriction, yes / no
Radiographic response (RR) - Diffusion restriction | 3 months
  Diffusion restriction, yes / no
Radiographic response (RR) - Diffusion restriction | 6 months
  Diffusion restriction, yes / no

SECONDARY OUTCOMES:
Vestibular Function | Baseline
  Video-Head Impulse Test (vHIT)
Vestibular Function | 3 months
  Video-Head Impulse Test (vHIT)
Vestibular Function | 6 months
  Video-Head Impulse Test (vHIT)
Vestibular Function | Baseline
  cervical Vestibular Evoked Myogenic Potential (cVEMP) test
Vestibular Function | 3 months
  cervical Vestibular Evoked Myogenic Potential (cVEMP) test
Vestibular Function | 6 months
  cervical Vestibular Evoked Myogenic Potential (cVEMP) test
Vestibular Function | Baseline
  Caloric test
Vestibular Function | 3 months
  Caloric test
Vestibular Function | 6 months
  Caloric test
Patient reported outcome measures (PROM) | Baseline
  Questionnaire on Quality of Life, and presence of symptoms
Patient reported outcome measures (PROM) | 3 months
  Questionnaire on Quality of Life, and presence of symptoms
Patient reported outcome measures (PROM) | 6 months
  Questionnaire on Quality of Life, and presence of symptoms
Physical examination | Baseline
  General neurological examination is performed to assess if the patient has neurological symptoms, if any. The examination is done according to standard clinical care and has a descriptive nature. Cranial nerve (dys)function, including House Brackmann scale for the facial nerve (n. VII) and trigeminal nerve function (n. V), including presence of neuralgia and hypoesthesia, are described in more detail.
Physical examination | 3 months
  General neurological examination is performed to assess if the patient has neurological symptoms, if any. The examination is done according to standard clinical care and has a descriptive nature. Cranial nerve (dys)function, including House Brackmann scale for the facial nerve (n. VII) and trigeminal nerve function (n. V), including presence of neuralgia and hypoesthesia, are described in more detail.
Physical examination | 6 months
  General neurological examination is performed to assess if the patient has neurological symptoms, if any. The examination is done according to standard clinical care and has a descriptive nature. Cranial nerve (dys)function, including House Brackmann scale for the facial nerve (n. VII) and trigeminal nerve function (n. V), including presence of neuralgia and hypoesthesia, are described in more detail.
Renal function | Baseline
  Creatinine clearance (CrCl), eGFR (mL/minute, ref. >90)
Renal function | 3 months
  Creatinine clearance (mmol/L), eGFR (mL/minute)
Renal function | 6 months
  Creatinine clearance (mmol/L), eGFR (mL/minute)

CONTACTS AND LOCATIONS:
Overall Officials: Hans AJ Gelderblom, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided